CLINICAL TRIAL: NCT06763328
Title: Metformin (Dimethylbiguanide) and Insulin Resistance in Women Completing Neoadjuvant and/or Adjuvant Cytotoxic Treatment of Stage I-III Breast Cancer
Brief Title: Metformin for the Treatment of Insulin Resistance in Women With Stage I-III Breast Cancer Completing Chemotherapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24363; NCI-2024-10402 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24363 (Other: City of Hope Medical Center); P30CA033572 (NIH); U54CA285116 (NIH)
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Invasive Breast Carcinoma
MeSH Terms: interventions — Specimen Handling; Early Intervention, Educational; Educational Status; Methods; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (standard of care, metformin) (Experimental): Patients receive standard of care healthy diet and exercise handouts and extended release metformin PO QD for 12 months in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Other: Educational Intervention; Drug: Extended Release Metformin Hydrochloride; Other: Questionnaire Administration
- Arm II (standard of care) (Active Comparator): Patients receive standard of care healthy diet and exercise handouts on study. Additionally, patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Other: Educational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Educational Intervention — Receive standard of care healthy diet and exercise handouts
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Drug: Extended Release Metformin Hydrochloride — Given PO
  Other Names: ER Metformin Hydrochloride; Extended-release Metformin Hydrochloride; Glucophage XR; Glumetza; Metformin Hydrochloride Extended Release
  Arms: Arm I (standard of care, metformin)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial evaluates how often women develop insulin resistance and type-2 diabetes and compares metformin with usual care to usual care alone in treating insulin resistance in women with stage I-III breast cancer after chemotherapy. Insulin resistance occurs when cells stop responding to insulin and is a risk factor for developing diabetes and heart disease. Higher levels of insulin have been shown to be associated with aggressive breast cancer. Metformin hydrochloride decreases the amount of glucose (a type of sugar) released into the bloodstream from the liver and increases the body's use of the glucose. Metformin as well as standard of care diet and exercise education is known to lower blood sugar. However, chemotherapy may accelerate metabolic disorders, such as high blood sugar, and the impact of metformin in these breast cancer survivors is not known. Giving metformin with usual care may be more effective than usual care alone in preventing or reversing insulin resistance in women with stage I-III breast cancer after chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if extended release metformin hydrochloride (metformin) can normalize glycosylated hemoglobin (HgbA1c) (< 5.7%) for women breast cancer survivors with HgbA1c between 5.7-6.4%.

EXPLORATORY OBJECTIVES:

I. To investigate whether metformin treatment of insulin resistance (versus standard of care alone) alters epigenetic changes (chromatin acetylation, chromatin opening, and methylation) and the level of inflammatory cytokines. (Pilot) II. To investigate whether normalization of HgbA1c alters epigenetic changes (chromatin acetylation, chromatin opening, and methylation) and the level of inflammatory cytokines. (Pilot)

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard of care healthy diet and exercise handouts and extended release metformin orally (PO) once daily (QD) for 12 months in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection throughout the study.

ARM II: Patients receive standard of care healthy diet and exercise handouts on study. Additionally, patients undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days and in 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Agreement to allow lab draw of approximately 26 mL of blood (less than 3 tablespoons)

  * To check blood counts, organ function and disease at baseline and 12 months
  * Clinical labs at baseline, 3 months, 6 months,12 months, and 24 months
  * Research labs at baseline, 6 months,12 months, and 24 months
* Age: ≥ 18 years
* Female sex assigned at birth
* Ability to read and understand English or Spanish for questionnaires
* Diagnosis of estrogen receptor (ER)-negative /HER2-wild type or -amplified invasive mammary carcinoma stages I-III
* Receive systemic treatment for breast cancer treatment
* Completed treatment for stage 1-3 breast cancer within 90 days to 5 years and are disease free
* Women who receive drugs for weight loss - e.g. semaglutide - prior to diagnosis are eligible for this protocol and can continue the drug during the intervention

Exclusion Criteria:

* Currently taking metformin or any other oral antidiabetic medications. Weight loss medications are permitted - e.g. semaglutide
* Taking tamoxifen or aromatase inhibitor
* Contraindication to metformin prevention such as acute hypersensitivity or allergic reaction to metformin
* Participants with acute or chronic renal insufficiency (a glomerular filtration rate [GFR] < 30 mL/min/1.73m^2) or those with acute renal insufficiency of any severity due to hepato-renal syndrome or in the peri-operative liver transplantation period
* Previously diagnosed type 1 or type 2 diabetes
* Patients pregnant or within 1 year of pregnancy and completion of lactation (pregnancy tests are standard of care [SOC] for initiation of chemotherapy)
* Other active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* An employee who is under the direct/indirect supervision of the principal investigator (PI)/a co-investigator/the study manager and/or a direct study team member
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2029-06-16 (Estimated); Study Completion 2029-06-16 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c (Hgb A1c) normalization | Up to 12 months
  Will be defined as Hgb A1c < 5.7%. Will be compared across groups (metformin + standard of care/usual medical care versus standard of care/usual medical care alone) using chi-square statistics. Data will be summarized using counts and percentages.

SECONDARY OUTCOMES:
HgbA1c normalization | At 3, 6, 12 and 24 months
  Will compare HgbA1c normalization as well as pairwise t-tests across treatment groups to examine the magnitude of change in HgbA1c.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria L Seewaldt, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California-Riverside, Riverside, California